CLINICAL TRIAL: NCT07346378
Title: Clinical Study on the Safety and Efficacy of Temporal Interference Stimulation in the Treatment of Post-Stroke Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Principal Investigator, hupanpan, Department of Neurology, The First Affiliated Hospital of Anhui Medical University,Hefei,China, The First Affiliated Hospital of Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHMU-TI-PSA
Record Dates: First submitted 2025-12-18; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Post-stroke Aphasia
MeSH Terms: interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Temporal interference stimulation (TI) will be applied for treatment; the current frequencies will be set at 1400 Hz and 1430 Hz; stimulation duration will be 30 minutes per session, once daily for 10 consecutive days.During the stimulation, they underwent standardized speech and language therapy (SLT) simultaneously.
  Interventions: Other: temporal interference stimulation; Behavioral: speech and language therapy
- sham stimulation (Sham Comparator): In the sham condition, TI was delivered only during the ramp-up and ramp-down periods (15 and 15 s); no current was delivered during the 30-minute intervention. Participants will receive sham TI once daily for 10 days. During the stimulation, they underwent standardized speech and language therapy (SLT) simultaneously.
  Interventions: Other: temporal interference stimulation; Behavioral: speech and language therapy

INTERVENTIONS:
Other: temporal interference stimulation — The envelope frequency of the TIS employed is set at 30 Hz, while the current frequencies are planned to be 1400 Hz and 1430 Hz. Due to individual variability in sensitivity to TIS, we intend to make necessary adjustments to the stimulation frequency or duration during the treatment process. For the continuous stimulation mode of TIS, the protocol follows the post-operative control consensus from Chinese experts in deep brain stimulation for neurological disorders. Electrode placement adheres to the international 10-10 EEG electrode system, with stimulation parameters (electrode positions and current parameters) determined based on the TIS optimization method proposed by the project team. The constraints are as follows: the total current across all electrodes must be less than 10 mA, and the maximum current for any single electrode is limited to 2.5 mA. The ramp-up time for stimulation is set at 30 seconds. The stimulation target for this project is based on MRI localization.
Behavioral: speech and language therapy — Speech and Language Therapy (SLT) was conducted by a certified Speech-Language Pathologist (SLP), providing standardized language rehabilitation for 40 minutes daily, which included 30 minutes of SLT synchronized with TI. Based on the results of the patients' language assessments, the SLP developed and implemented an individualized rehabilitation treatment plan. The primary rehabilitation methodologies included articulation exercises, phoneme stimulation, Schuell stimulation therapy, melodic intonation therapy, object naming exercises, word reading practice, and situational conversation practice.

SUMMARY:
Neurological disorders encompass a wide variety of diseases, including congenital and neurodevelopmental disorders, cerebrovascular and neurodegenerative diseases, nervous system infections, neuroimmune diseases, neuromuscular or peripheral nervous system disorders, traumatic injuries, and tumor-related neurological conditions, with diverse symptomatic manifestations. The etiology, symptoms, and disease courses of these disorders vary significantly, severely impacting human health and social development, and have become a critical global public health issue. Some neurological disorders can lead to lifelong disability or high mortality rates, while others remain poorly understood, lacking effective treatments or cures.

Post-stroke aphasia (PSA) is an acquired language impairment caused by ischemic or hemorrhagic injuries to the central nervous system. Its clinical manifestations are diverse, potentially affecting spontaneous speech, auditory comprehension, repetition, naming, reading, and writing abilities, among other aspects. Statistics indicate that over 16 million people worldwide suffer from stroke each year, with approximately 38% of survivors experiencing aphasia. The prognosis for this condition is concerning, as more than 40% of patients still exhibit significant language impairments one year after the stroke, with some even facing lifelong effects. The large patient population, significant communication barriers, and poor prognosis severely diminish patients' quality of life, significantly increasing their risk of emotional disorders such as depression and social isolation. This poses a substantial challenge to family caregiving and public health systems. Therefore, the development of non-invasive and effective novel therapeutic approaches holds substantial scientific and societal importance.

Temporal interference stimulation (TI) technology represents a breakthrough in achieving non-invasive deep brain stimulation. This technology is based on the interference phenomenon, utilizing two pairs of surface electrodes to simultaneously apply sinusoidal wave stimuli at 2 kHz and 2.01 kHz. Two cortical regions are exposed to electric fields of 2 kHz or 2.01 kHz, and an interference electric field is generated in the brain region where these two fields overlap, with its envelope oscillating at 10 Hz. This technology has already been applied in the treatment of conditions such as depression, Parkinson's disease, and disorders of consciousness. The primary objective of this study is to explore the effects of TI intervention on deep brain regions, particularly on motor and non-motor related brain networks and functions in patients with neurological disorders, especially post-stroke aphasia. This research aims to provide a potential new approach for improving the clinical symptoms of these patients.

DETAILED DESCRIPTION:
This study plans to recruit 40 patients with neurological disorders and randomly assign them to either a real stimulation treatment group or a sham stimulation treatment group (20 patients per group). The real stimulation treatment group will receive treatment using Temporal Interference Stimulation (TIS) technology. The current frequencies are intended to be 1400 Hz and 1430 Hz. The stimulation duration is 30 minutes; administered once daily for 10 consecutive days. The control group will receive sham stimulation. The sham stimulation group will have the same electrode placement, current intensity, and frequency settings as the TIS group, but without eliciting physiological effects. Randomization will be performed to blind both the patients and the assessors. The order of stimulation targets will be randomized between subjects, while the order of stimulation targets for the same subject will remain consistent throughout the treatment course. Treatment will be administered for 10 consecutive days. Both groups will receive either real or sham stimulation paired simultaneously with standard Speech and Language Therapy (SLT).The observation indicators will be the changes in scores from baseline to post-treatment and follow-up on the following assessments: Western Aphasia Battery (WAB, including fluency and information content), Aphasia Battery of Chinese (ABC,comprising spontaneous speech, auditory comprehension, repetition, naming, reading, writing, structural and spatial functions, application and calculation), Verbal Fluency Test (VFT), Language Assessment Manual (Including True Word Auditory Repetition, Picture Naming, Non-Word Auditory Repetition, Word Reading, Verb-Noun-Picture Matching, Writing), Mini-Mental State Examination (MMSE), Montreal Cognitive Assessment (MoCA), Activities of Daily Living (ADL) scale, Hamilton Depression Rating Scale (HAMD), Hamilton Anxiety Rating Scale (HAMA), Brunnstrom stages of stroke recovery, and simplified Fugl-Meyer Assessment of motor function (FMA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with post-stroke aphasia;
* Right-handed;
* Native Chinese speaker with comprehension of Mandarin;
* Aged 18-80 years;
* Complete relevant assessment and imaging data;
* Informed consent obtained from the patient and their family.

Exclusion Criteria:

* Cerebellar involvement in the stroke lesion, and incomplete scanning of cerebellar structures;
* Severe dysarthria;
* Concurrent epilepsy with occasional seizures;
* Implanted pacemaker or deep brain stimulator;
* History of brain tissue resection for prior lesions such as brain tumours or brain abscesses;
* Other severe psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Aphasia Battery of Chinese (ABC,comprising spontaneous speech, auditory comprehension, repetition, naming, reading, writing, structural and spatial functions, application and calculation) | Baseline;10 days; one-month follow-up
  Language deficit was assessed by the same professional language therapist using the Aphasia Battery of Chinese (ABC). The multidimensional test contains four subtypes, including spontaneous speech (semi-standardized interview, assessment of the fluency, and information of speech; total score 20 points), auditory comprehension (yes or no question, auditory picture matching task, and verbal instruction; total score 230 points), repetition (words and sentences; total score 100 points), naming (simple objects, colors, pictures, and situations; total score 80 points), structural and spatial functions (draw the picture; total score 19 points), application (total score30 points), and calculation (total score20 points). The combined score is used to calculate an aphasia quotient (AQ) reflecting the overall severity of language impairment. Patients with AQ below 93.8 points were considered as aphasic.
Verbal fluency test (VFT) | Baseline;10 days; one-month follow-up
  The Verbal Fluency Test (VFT) is a cognitive assessment tool used to evaluate language production and executive function, where individuals generate words based on specific criteria within a one-minute timeframe. The total score reflects the number of acceptable words produced: for phonemic fluency, participants generate words starting with a specific letter, while for semantic fluency, they list words belonging to a designated category; scores typically range from 0 to 60, with higher scores indicating better verbal fluency and cognitive function.
Western Aphasia Battery (WAB, including fluency and information content) | Baseline;10 days; one-month follow-up
  The Western Aphasia Battery (WAB) is a comprehensive assessment tool designed to evaluate language abilities in individuals with aphasia, measuring various aspects of verbal communication, including fluency and information content. The total score for the WAB ranges from 0 to 100, with higher scores indicating better overall language function and less severe aphasia. Specifically, fluency assesses the ease and flow of speech, while information content evaluates the meaningfulness and relevance of the verbal output.

SECONDARY OUTCOMES:
Language Assessment Manual (Including True Word Auditory Repetition, Picture Naming, Non-Word Auditory Repetition, Word Reading, Verb-Noun-Picture Matching, and Writing) | Baseline;10 days; one-month follow-up
  The Language Assessment Manual, developed by the University of Hong Kong, is a comprehensive evaluation tool that assesses various aspects of language function, including True Word Auditory Repetition, Picture Naming, Non-Word Auditory Repetition, Word Reading, Verb-Noun-Picture Matching, and Writing. Each dimension of the assessment contributes to an overall score, with True Word Auditory Repetition, Picture Naming, Non-Word Auditory Repetition, and Word Reading each contributing up to 10 points; Verb-Noun-Picture Matching contributing up to 15 points; and the Writing component contributing a maximum of 15 points, resulting in a total possible score of 70. Higher scores indicate better language abilities, reflecting enhanced communication skills across the assessed modalities. This manual serves as a vital resource in both clinical and research settings, providing valuable insights into the linguistic capabilities of individuals with language impairments, facilitating tailored interv
Mini Mental State Examination (MMSE) | Baseline;10 days;one-month follow-up
  The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answe he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better.
Montreal Cognitive Assessment (MoCA) | Baseline;10 days; one-month follow-up
  The Montreal Cognitive Assessment (MoCA) is a widely utilized cognitive evaluation tool designed to assist in the identification of mild cognitive impairment. The tool is scored out of a total of 30 points, with assessment divided across several dimensions, including attention (5 points), memory (5 points), language (6 points), visuospatial abilities (5 points), executive function (5 points), and abstraction (2 points), alongside orientation (6 points). In this scale, higher scores indicate better cognitive functioning, with a scoring range from 0 (indicating severe cognitive impairment) to 30 (reflecting normal cognitive function). This assessment provides clinicians with a convenient and effective means of evaluating a patient's cognitive status, thereby facilitating further diagnostic and therapeutic interventions.
Brunnsrom stages of motor recovery | Baseline;10 days; one-month follow-up
  The Brunnstrom Stages of Motor Recovery is an assessment tool specifically designed to evaluate the recovery of motor function in stroke patients, delineating the progression of motor recovery through seven distinct stages. Each stage reflects the functional abilities and associated neurological recovery. The scoring system within the Brunnstrom approach does not assign a numerical total score as other standardized assessments do; instead, it categorizes patient recovery into stages ranging from Stage I (flaccidity, no voluntary movement) to Stage VII (normal motor function). As patients progress from Stage I to Stage VII, they demonstrate increasing levels of voluntary control, coordination, and skill in movement execution, indicating better motor recovery. Thus, while there is no fixed scoring range, advancement through the seven stages signifies improving motor function and recovery post-stroke, serving as a crucial framework for clinicians to guide rehabilitation interventions.
Fugl-Meyer Assessment Scale (FMA) | Baseline;10 days; one-month follow-up
  The Fugl-Meyer Assessment (FMA) is a comprehensive and widely used evaluation tool for assessing motor function, sensory function, balance, and joint function in individuals who have experienced a stroke or other neurological conditions. The total score for the FMA is 226 points, which is divided across several domains: motor function (upper extremity) scores a maximum of 66 points, motor function (lower extremity) scores a maximum of 34 points, sensory function scores a maximum of 24 points, balance scores a maximum of 14 points, and joint function and pain scores 8 points. Additionally, there is a reflex assessment with a maximum of 14 points, contributing to the overall score. Higher scores indicate better motor and sensory recovery, with the minimum score being 0, representing complete functional loss. This assessment serves as a vital tool for clinicians to gauge recovery progress and plan appropriate rehabilitation interventions for patients following a stroke or similar injury.
Hamilton Anxiety Rating Scale (HAMA) | Baseline;10 days; one-month follow-up
  The Hamilton Anxiety Rating Scale (HAMA) is a clinician-administered assessment tool used to quantify the severity of anxiety symptoms in patients. The scale comprises 14 items, each focusing on different dimensions of anxiety, including psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical symptoms). The total score ranges from 0 to 56, with higher scores indicating greater severity of anxiety symptoms: a score of 0-17 represents mild anxiety, 18-24 indicates moderate anxiety, and 25-56 signifies severe anxiety. The HAM-A provides a structured method for clinicians to evaluate anxiety levels over time, facilitating treatment planning and monitoring of the patient's response to therapeutic interventions.
Hamilton Depression Rating Scale (HAMD) | Baseline;10 days; one-month follow-up
  The Hamilton Depression Rating Scale (HAMD) is a widely used clinician-administered tool designed to assess the severity of depression in individuals. The total score can vary depending on the specific version of the scale used, with the most common version containing 17 items, yielding a total score ranging from 0 to 54, where higher scores reflect more severe depressive symptoms. The scale covers several dimensions of depression, including mood, guilt, suicide ideation, insomnia, work and activities, psychomotor retardation, agitation, anxiety, weight loss, insight, and somatic symptoms, with each item scored on a scale of 0 to 4 or 0 to 2, depending on the symptom's severity. A score of 0-7 typically indicates no depression, 8-13 indicates mild depression, 14-18 indicates moderate depression, and scores above 18 suggest severe depression. The HAMD is essential for clinicians to evaluate depressive severity, facilitate treatment planning, and monitor changes in a patient's depressiv
MRI measures | Baseline;10 days; one-month follow-up
  Multimodal magnetic resonance data were acquired, including structural phase magnetic resonance and rest state magnetic resonance.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
Six months after the end of the study, it can be obtained via email with the researcher's consent.